CLINICAL TRIAL: NCT06334432
Title: A Phase 1/2, First-in-Human, Safety and Efficacy Study of NUV-1511 in Adult Patients With Advanced Solid Tumors
Brief Title: Safety and Efficacy Study of NUV-1511 in Adult Patients With Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nuvation Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NUV-1511-01
Record Dates: First submitted 2024-02-12; First posted 2024-03-28 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumor; HER2-negative Breast Cancer; Metastatic Castration-resistant Prostate Cancer (mCRPC); Pancreatic Cancer; Platinum-resistant Ovarian Cancer (PROC)
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Phase 1: Schedule A (Other): Schedule A evaluating escalating dose levels of NUV-1511
  Interventions: Drug: NUV-1511
- Phase 1: Schedule B (Other): Schedule B evaluating escalating dose levels of NUV-1511
  Interventions: Drug: NUV-1511
- Phase 2: Tumor Type 1 (Experimental): Tumor type to be selected after Phase 1. Dose Schedules A and B to be further evaluated.
  Interventions: Drug: NUV-1511
- Phase 2: Tumor Type 2 (Experimental): Tumor type to be selected after Phase 1. Dose level and schedule to be selected after identification of the recommended phase 2 dose (RP2D) in Phase 1.
  Interventions: Drug: NUV-1511
- Phase 2: All comers (Experimental): All tumor types allowed per protocol. Dose level and schedule to be selected after identification of the recommended phase 2 dose (RP2D) in Phase 1.
  Interventions: Drug: NUV-1511

INTERVENTIONS:
Drug: NUV-1511 — Novel small molecule

SUMMARY:
NUV-1511-01 is a first-in human, open- label, Phase 1/2 to evaluate the safety and efficacy of NUV-1511 in patients with advanced solid tumors. The Phase 1 portion include patients with advanced solid tumors and is designed to determine the safety and the tolerability of doses of NUV-1511. In Phase 2, NUV-1511 will be given to determine the efficacy of patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Phase 1 Dose Escalation cohorts, Phase 1 Backfill cohorts, and Phase 2 Tumor Type-Specific cohort(s): must meet one of the following criteria:
* HER2- metastatic breast cancer:

  1. Hormone refractory hormone receptor positive metastatic breast cancer with progression on or after treatment with CDK4/6 inhibitor plus at least one line of systemic chemotherapy in the advanced setting
  2. Triple negative metastatic breast cancer with progression after at one line of systemic chemotherapy in the advanced setting.
* Patients with advanced solid tumors that progressed on or following treatment with Enhertu and/or Trodelvy per label
* mCRPC: Histologically confirmed, metastatic castration resistant adenocarcinoma of the prostate

  1. May have received up to 2 prior chemotherapies in mCRPC setting
  2. Prior therapy with PARP (poly-ADP ribose polymerase) inhibitor, PLUVICTO, Radium-223, or Provenge is allowed
* Pancreatic cancer: PDAC (pancreatic ductal adenocarcinoma) with progression on or after treatment with at least one line of systemic chemotherapy in the advanced setting.
* PROC: Histologically or cytologically confirmed platinum-resistant high-grade serous ovarian, fallopian, or primary peritoneal cancer;
* Phase 1 Dose Escalation cohorts, Phase 1 Backfill cohorts, and Phase 2 Tumor Type-Specific cohorts (except mCRPC; see inclusion criterion 2 above): must have measurable disease per RECIST 1.1
* Phase 2 All Comers cohort: Patients with advanced solid tumors that have progressed during or after treatment with approved therapies or for whom there is no standard effective therapy available.
* Adequate bone marrow and organ function.
* Provide informed consent, which includes compliance with protocol-specified requirements and restrictions

Exclusion Criteria:

* Chemotherapy, hormonal therapy (with the exception of ongoing luteinizing hormone-releasing hormone analogs in male patients and premenopausal females), radiation therapy, or biological anticancer therapy within 14 days before the first dose of study treatment
* Treatment with an investigational agent for any indication within 14 days before the first dose of study treatment for non-myelosuppressive agent, or within 21 days or <5 half-lives before the first dose of study treatment, whichever is longer, for a myelosuppressive agent
* Ongoing or active infection requiring systemic therapy, or an infection requiring hospitalization or intravenous therapy within 2 weeks before the first dose of study treatment
* Resting left ventricular ejection fraction (LVEF) of <50% obtained by echocardiography or multigated acquisition scan (MUGA)
* History of significant cardiac disease, including myocardial infarction, New York Heart Association Class II/III/IV heart failure, unstable angina, unstable cardiac arrhythmias (eg, ventricular tachycardia, ventricular fibrillation), syncope of cardiovascular etiology, or cardiac arrest:
* Known immunosuppressive disease or active systemic autoimmune disease such as systemic lupus erythematosus, human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV) infections not currently controlled by current disease-specific therapy. The following exceptions apply:
* Major surgical procedure within 2 weeks before the first dose of study treatment, or an anticipated need for major surgery during the course of the study
* Other cancer within 2 years before the first dose of study treatment with metastatic or local recurrence potential that could negatively impact survival and/or potentially confound tumor response assessments. Patients with a history of other cancers in the past 2 years should be discussed with the Medical Monitor.
* Female patients who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 466 (Estimated)
Dates: Start 2024-03-14 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Assess safety and tolerability of NUV-1511 in advanced solid tumors | First 28 days of dosing (DLT evaluation period)
  Number of patients with dose limiting toxicities, treatment emergent adverse events (TEAE) and serious adverse events (SAE) and laboratory abnormalities
Phase 1: Identify recommended dosing schedule(s) and corresponding Phase 2 dose(s) (RP2D(s)) | First 28 days of dosing (DLT evaluation period)
  Number of patients with DLTs, TEAEs and SAEs and laboratory abnormalities
Phase 2: Evaluate the efficacy of NUV-1511 in advanced solid tumors and selected tumor type(s) | From date of enrollment to date of disease progression, withdrawal of consent, or initiation of subsequent anticancer treatment or up to a period of 5 years, whichever occurs first
  Efficacy measures may include tumor assessments, as assessed by CT scans, PET/CT, whole body bone scan and MRI
Phase 2: Confirm the optimal NUV-1511 dose level/schedule for further development | Periodic efficacy assessments from date of enrollment to date of disease progression, withdrawal of consent, or initiation of subsequent anticancer treatment or up to a period of 5 years, whichever occurs first
  Overall response rate per RECIST 1.1 (Composite response rate for mCRPC patients only, if enrolled in Phase 2)
Phase 2: Confirm the optimal NUV-1511 target tumor types for further development | Periodic efficacy assessments from date of enrollment to date of disease progression, withdrawal of consent, or initiation of subsequent anticancer treatment or up to a period of 5 years, whichever occurs first
  Overall response rate per RECIST 1.1 (Composite response rate for mCRPC patients only, if enrolled in Phase 2)

SECONDARY OUTCOMES:
Phase 1: Explore preliminary efficacy of NUV-1511 | From date of enrollment to date of disease progression, withdrawal of consent, or initiation of subsequent anticancer treatment or up to a period of 5 years, whichever occurs first
  Overall response rate and duration of response per RECIST 1.1. Efficacy measures may include tumor assessments, as assessed by CT scans, PET/CT, whole body bone scan and MRI.
Phase 1: Explore preliminary efficacy of NUV-1511 | From date of enrollment to date of disease progression, withdrawal of consent, or initiation of subsequent anticancer treatment or up to a period of 5 years, whichever occurs first
  Overall response rate and duration of response per composite response rate (for mCRPC). Efficacy measures may include tumor assessments, as assessed by CT scans, PET/CT, whole body bone scan and MRI.
Phase 1: Explore preliminary efficacy of NUV-1511 | From date of enrollment to date of disease progression, withdrawal of consent, or initiation of subsequent anticancer treatment or up to a period of 5 years, whichever occurs first
  Overall response rate and duration of response per response rates in specific disease markers. Efficacy measures may include tumor assessments, as assessed by CT scans, PET/CT, whole body bone scan and MRI.
Characterize the PK profile of NUV-1511 | Periodic PK sample collection from date of enrollment to date of disease progression, withdrawal of consent, or initiation of subsequent anticancer treatment or up to a period of 5 years, whichever occurs first.
  Parameters include, but not limited to, maximum observed plasma concentration (Cmax)
Characterize the PK profile of NUV-1511 | Periodic PK sample collection from date of enrollment to date of disease progression, withdrawal of consent, or initiation of subsequent anticancer treatment or up to a period of 5 years, whichever occurs first.
  Parameters include, but not limited to, area under the plasma concentration-time curve (AUC)
Phase 2: Further evaluate the safety and efficacy of NUV-1511 | Ongoing monitoring of safety and efficacy from date of enrollment to date of disease progression, withdrawal of consent, or initiation of subsequent anticancer treatment or up to a period of 5 years, whichever occurs first
  Incidence of TEAEs and SAEs
Phase 2: Further evaluate the safety and efficacy of NUV-1511 | Ongoing monitoring of safety and efficacy from date of enrollment to date of disease progression, withdrawal of consent, or initiation of subsequent anticancer treatment or up to a period of 5 years, whichever occurs first
  Laboratory abnormalities
Phase 2: Further evaluate the safety and efficacy of NUV-1511 | Ongoing monitoring of safety and efficacy from date of enrollment to date of disease progression, withdrawal of consent, or initiation of subsequent anticancer treatment or up to a period of 5 years, whichever occurs first
  Duration of response
Phase 2: Further evaluate the safety and efficacy of NUV-1511 | Ongoing monitoring of safety and efficacy from date of enrollment to date of disease progression, withdrawal of consent, or initiation of subsequent anticancer treatment or up to a period of 5 years, whichever occurs first
  Clinical best response
Phase 2: Further evaluate the safety and efficacy of NUV-1511 | Ongoing monitoring of safety and efficacy from date of enrollment to date of disease progression, withdrawal of consent, or initiation of subsequent anticancer treatment or up to a period of 5 years, whichever occurs first
  Progression free survival
Phase 2: Further evaluate the safety and efficacy of NUV-1511 | Ongoing monitoring of safety and efficacy from date of enrollment to date of disease progression, withdrawal of consent, or initiation of subsequent anticancer treatment or up to a period of 5 years, whichever occurs first
  Overall survival
Phase 2: Further evaluate the safety and efficacy of NUV-1511 | Ongoing monitoring of safety and efficacy from date of enrollment to date of disease progression, withdrawal of consent, or initiation of subsequent anticancer treatment or up to a period of 5 years, whichever occurs first
  PK exposure-response modeling, which includes measuring plasma concentration versus overall response rate
Phase 2: Further evaluate the safety and efficacy of NUV-1511 | Ongoing monitoring of safety and efficacy from date of enrollment to date of disease progression, withdrawal of consent, or initiation of subsequent anticancer treatment or up to a period of 5 years, whichever occurs first
  PK exposure-response modeling, which includes measuring plasma concentration versus progression free survival
Phase 2: Further evaluate the safety and efficacy of NUV-1511 | Ongoing monitoring of safety and efficacy from date of enrollment to date of disease progression, withdrawal of consent, or initiation of subsequent anticancer treatment or up to a period of 5 years, whichever occurs first
  PK exposure-response modeling, which includes measuring plasma concentration versus treatment emergent adverse events and serious adverse events.
Phase 2: Further evaluate the safety and efficacy of NUV-1511 | Ongoing monitoring of safety and efficacy from date of enrollment to date of disease progression, withdrawal of consent, or initiation of subsequent anticancer treatment or up to a period of 5 years, whichever occurs first
  Response rates in disease-specific markers

OTHER OUTCOMES:
Phase 1 and Phase 2: Evaluate biomarkers potentially related to NUV-1511 anti-tumor activity via ctDNA and tumor tissue analysis | Ongoing monitoring of safety and efficacy from date of enrollment to date of disease progression, withdrawal of consent, or initiation of subsequent anticancer treatment or up to a period of 5 years, whichever occurs first
  Blood sample for exploratory analysis of circulating DNA
Phase 1 and Phase 2: Evaluate biomarkers potentially related to NUV-1511 anti-tumor activity via ctDNA and tumor tissue analysis | Ongoing monitoring of safety and efficacy from date of enrollment to date of disease progression, withdrawal of consent, or initiation of subsequent anticancer treatment or up to a period of 5 years, whichever occurs first
  Blood sample for exploratory analysis of gene expression (including that of hormone receptors and efflux transporters)
Phase 1 and Phase 2: Evaluate biomarkers potentially related to NUV-1511 anti-tumor activity | Ongoing monitoring of safety and efficacy from date of enrollment to date of disease progression, withdrawal of consent, or initiation of subsequent anticancer treatment or up to a period of 5 years, whichever occurs first
  Tumor biopsy for exploratory analysis of tumor genome
Phase 1 and Phase 2: Evaluate biomarkers potentially related to NUV-1511 anti-tumor activity | Ongoing monitoring of safety and efficacy from date of enrollment to date of disease progression, withdrawal of consent, or initiation of subsequent anticancer treatment or up to a period of 5 years, whichever occurs first
  Tumor biopsy for exploratory analysis of epigenome
Phase 1 and Phase 2: Evaluate biomarkers potentially related to NUV-1511 anti-tumor activity | Ongoing monitoring of safety and efficacy from date of enrollment to date of disease progression, withdrawal of consent, or initiation of subsequent anticancer treatment or up to a period of 5 years, whichever occurs first
  Tumor biopsy for exploratory analysis of gene expression
Phase 1 and Phase 2: Explore pharmacogenetic profiling that may be potentially predictive of NUV-1511 antitumor activity or toxicity | Blood and tumor biopsy collection at the time of enrollment
  Identification of genetic factors that predict toxicity
Phase 1 and Phase 2: Explore pharmacogenetic profiling that may be potentially predictive of NUV-1511 antitumor activity or toxicity | Blood and tumor biopsy collection at the time of enrollment
  Identification of genetic factors that predict anti-tumor activity
Phase 1 and Phase 2: Explore pharmacogenetic profiling that may be potentially predictive of NUV-1511 antitumor activity or toxicity | Blood and tumor biopsy collection at the time of enrollment
  Identification of genetic factors that predict metabolism of NUV-1511
Evaluate drug exposure-response relationship | Periodic PK sample collection through disease progression, withdrawal of consent, or initiation of subsequent anticancer treatment or up to a period of 5 years, whichever occurs first
  PK exposure response modeling which includes measuring PK exposure versus efficacy
Evaluate drug exposure-response relationship | Periodic PK sample collection through disease progression, withdrawal of consent, or initiation of subsequent anticancer treatment or up to a period of 5 years, whichever occurs first
  PK exposure response modeling which includes measuring PK exposure versus safety

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Karmanos Cancer Center, Detroit, Michigan
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Carolina BioOncology Institute, Huntersville, North Carolina
  - NEXT Oncology, Irving, Texas
  - START Mountain, Salt Lake City, Utah
  - NEXT Oncology, Fairfax, Virginia
  - Fred Hutchinson, Seattle, Washington